CLINICAL TRIAL: NCT02058342
Title: Family-based Exercise Intervention for Children and Adolescents With Prader-Willi Syndrome
Brief Title: Family-based Intervention for Youth With Prader-Willi Syndrome: The Active Play at Home Study
Acronym: APAH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: California State University, Fullerton (Other)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSR-13-0142.54155; W81XWH-09-1-0682 (Other Grant/Funding Number: USAMRAA)
Record Dates: First submitted 2014-02-06; First posted 2014-02-10 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Prader Willi Syndrome; Childhood Obesity
Keywords: Prader Willi syndrome; Obesity; Childhood; Family; Interactive games; Playground games; Exercise routine
MeSH Terms: conditions — Prader-Willi Syndrome; Pediatric Obesity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Play at Home Intervention (Experimental): Participant parents in the intervention arm will receive: 1) Active Play at Home curriculum and equipment, 2) Training session on Active Play at Home curriculum, 3) counseling on physical activity scheduling, identification of barriers, motivational strategies, 4) phone calls to check on compliance and issues with doing the program at home
  Interventions: Behavioral: Active Play at Home
- Wait-listed control (No Intervention): Participants will attend the baseline visit to do baseline measurements but will not receive any materials related to the Active Play at Home curriculum and will also not be contacted by phone during the control 24 weeks. After they serve as control group, they will be provided with the opportunity to receive the intervention.

INTERVENTIONS:
Behavioral: Active Play at Home — The Active Play at Home (APAH) curriculum includes age-appropriate goal-oriented physical activities that combine playground and video games using the Nintendo Wii™ with exercises targeting: muscular strength and endurance, aerobic endurance, flexibility, balance, agility, and motor coordination. APAH was designed for children ages 8-11 without disability and ages 8-15 years with PWS. The playground games and interactive console-based games are to be performed twice weekly each. The activity is progressed from 25 to 45 minutes of moderate to vigorous physical activity throughout the 24 weeks period. Parents and children are trained to use the curriculum hands-on at baseline.
  Arms: Active Play at Home Intervention

SUMMARY:
Compared to other children, those with disability have additional challenges to being physically active. Prader-Willi Syndrome (PWS) is a genetic form of childhood obesity that is characterized by hypotonia, growth hormone deficiency, behavioral, and cognitive disability. In children, the low prevalence of PWS (1 in 10,000 to 15,000 live births) makes group-based physical activity (PA) interventions impossible. In contrast, the home environment presents a natural venue to establish a PA routine for this population. The present high prevalence of non-syndromal childhood obesity (one in four) and high physical inactivity rates, make alternative approaches to increasing PA in this population an area of high interest. Therefore, we have developed a 24-week home-based physical activity that could be suitable for children and adolescents ages 8-15 with PWS as well as obese children without PWS ages 8-11 years. It is hypothesized that: 1) an age-appropriate 24-week home-based PA intervention will increase PA levels in youth with PWS and without the syndrome but with obesity; 2) motor proficiency, central sensory reception and integration, and body composition will significantly improve in youth with and without PWS following completion of the home-based PA intervention and 3) physical activity self-efficacy and quality of life will increase significantly in youth with and without PWS who complete the home-based PA intervention. The study participants are 115 youth ages 8-15 y (45 with PWS and 70 without PWS but categorized as obese). The study utilizes a parallel design with the wait-listed control group receiving the intervention after serving as control. Participants are expected to complete the PA curriculum 4 days a week for six months including playground games 2 days a week and interactive console games 2 days a week. Parents are trained at baseline and then provided with a PA curriculum (Active Play at Home) and equipment to guide their implementation of the program at home. Measurements of children and parent dyads are assessed at baseline and at the end (week 24) of the intervention or control periods. Outcome measures include PA, body composition, motor proficiency, central sensory reception and integration (subsample of children only), quality of life and physical activity self-efficacy. PA intervention compliance is monitored using mail-in daily self-report checklists.

DETAILED DESCRIPTION:
Compared to other children, those with disability have additional challenges to being physically active. Prader-Willi Syndrome (PWS) is a genetic form of childhood obesity that is characterized by hypotonia, growth hormone deficiency, behavioral, and cognitive disability. In children, the low prevalence of PWS (1 in 10,000 to 15,000 live births) makes group-based physical activity (PA) interventions impossible. In contrast, the home environment presents a natural venue to establish a PA routine for this population. The present high prevalence of non-syndromal childhood obesity (one in four) and high physical inactivity rates, make alternative approaches to increasing PA in this population an area of high interest. Specifically, approaches that involve the family have been identified as possible areas where further research is needed. Therefore, we have developed a 24-week home-based physical activity that could be suitable for children and adolescents ages 8-15 with PWS as well as obese children without PWS ages 8-11 years. It is hypothesized that: 1) an age-appropriate 24-week home-based PA intervention will increase PA levels in youth with PWS and without the syndrome but with obesity; 2) motor proficiency, central sensory reception and integration, and body composition will significantly improve in youth with and without PWS following completion of the home-based PA intervention and 3) physical activity self-efficacy and quality of life will increase significantly in youth with and without PWS who complete the home-based PA intervention. The study participants are 115 youth ages 8-15 y (45 with PWS and 70 without PWS but categorized as obese). The study utilizes a parallel design with the wait-listed control group receiving the intervention after serving as control. Participants are expected to complete the PA curriculum 4 days a week for six months including playground games 2 days a week and interactive console games 2 days a week. Parents are trained at baseline and then provided with a PA curriculum (Active Play at Home) and equipment to guide their implementation of the program at home. Tips related to scheduling and coping with barriers to daily program implementation are also included. Throughout, parents are contacted by phone once a week (weeks 1-4) and then every other week to provide support in between visits. Measurements of children and parent dyads are assessed at baseline, at 12-weeks of receiving the intervention and at the end (week 24) of the intervention or control periods. PA intervention compliance is monitored using mail-in daily self-report checklists.

ELIGIBILITY:
Inclusion Criteria:

* Having Prader-Willi Syndrome and being between ages 8-15 years. PWS status will be documented by appropriate molecular and cytogenetic testing (i.e., chromosomes, florescence in situ hybridization [FISH] 15, DNA methylation, DNA polymorphism studies)
* Being obese and between ages 8-11 years. Obesity is defined as having a body fat percentage greater than the 95th percentile (McCarthy, H. D., Cole, T. J., Fry, T., Jebb, S. A., & Prentice, A. M. (2006). Body fat reference curves for children. International Journal of Obesity (Lond), 30(4), 598-602).

Exclusion Criteria:

* Obese children without Prader-Willi Syndrome currently on lipid-lowering medication, diabetes medications, or blood pressure medications.
* Being pregnant

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 115 (Estimated)
Dates: Start 2011-05; Primary Completion 2015-06 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Physical Activity | Baseline to 24 weeks
  PA level: This outcome will be measured using accelerometers which provide detailed information on the temporal patterns (duration, frequency, and intensity) of PA. Data are stored as acceleration counts and data can be downloaded to a personal computer. Youth will use the 4MB GT3X (Actigraph, Pensacola, FL) triaxial activity monitor at the hip for eight consecutive days. Participants should wear the monitor all day while they are awake and remove the monitor when they shower, bathe, swim, or do something that may get the monitor completely wet. The youth and parents will be asked to fill out a log of all the physical activities they engage in during the days they wear the accelerometer. The child will wear the accelerometer for eight days to capture two typical weekend days. Physical activity will be defined as minutes per day of Moderate to Vigorous Physical Activity. Accelerometry cut-points published by Evenson et al. will be used to determine MVPA.

SECONDARY OUTCOMES:
Body composition | Baseline to 24 weeks
  Percentage of body fat will be measured using dual x-ray absorptiometry (DXA) model Lunar Prodigy Advance Plus (GE Healthcare, Milwaukee, WI). For female participants who have had their first menses, a urine pregnancy test will be completed before conducting the DXA scan. A pregnancy test is required by law because the x-rays might be harmful to the fetuses. If the participant is pregnant, she will be excluded from the study as a major study outcome is body composition and the participant will experience changes in body composition because of pregnancy, thus invalidating the study findings.
Motor proficiency | Baseline to 24 weeks
  The Bruininks-Oseretsky Test of Motor Proficiency (BOTMP™-2) is used to evaluate overall motor proficiency. The BOTMP™-2 test measures fine manual control (fine motor precision and fine motor integration), manual coordination (manual dexterity and upper limb coordination), body coordination (bilateral coordination and balance), and strength and agility (running speed and agility and strength). This test also provides an overall motor proficiency score, as well as separate scores for the different domains of motor proficiency (Bruininks, R., Bruininks-Oseretsky test of motor proficiency: examiner's manual. 1978, MN: American Guidance Service). It is expected that significant improvements are demonstrated following completion of the PA intervention in the areas of upper limb coordination, bilateral coordination, balance, running speed, and agility and strength.
Sensory reception and motor integration | Baseline to 24 weeks
  Sensory reception and motor integration will be measured using The Sensory Organization Test. The SOT is designed to identify impairments in one or more of the three sensory systems (i.e., vision, somatosensory, vestibular) that contribute to standing balance. This test has been previously used with pediatric populations, with and without disabilities such as cerebral palsy. The test is comprised of six test conditions. This test will be administered only in a subsample of participants (30 with PWS and 55 with non-syndromal obesity).
Physical activity self-efficacy | Baseline to 24 weeks
  Self-efficacy for physical activity will be measured with an eight item questionnaire rated on a five point scale ranging from disagree a lot to agree a lot . This questionnaire was originally developed for use with children in fifth grade, but also validated with children in eighth grade. This questionnaire had a test-retest reliability of r= 0.84 over a period of two weeks. Additionally, the questionnaire had an internal consistency score of 0.88. Dishman, R.K., et al. Factorial invariance and latent mean structure of questionnaires measuring social-cognitive determinants of physical activity among black and white adolescent girls. Prev Med, 2002. 34(1): p. 100-8.
Quality of life | Baseline to 24 weeks
  will be measured using Pediatric Quality of Life Inventory (PedsQL™) to assess multidimensional constructs covering physical, emotional, mental, social, and behavioral components of well-being and function in youth (Varni, J.W., et al., The PedsQL 4.0 as a pediatric population health measure: feasibility, reliability, and validity. Ambul Pediatr, 2003. 3(6): p. 329-41)

OTHER OUTCOMES:
Anthropometrics | Baseline to 24 weeks
  Stature, measured to the nearest 0.1 cm using a wall-mounted stadiometer. Body mass, obtained to the nearest 0.1 kg following Third U.S. National Health and Nutrition Examination Survey procedures. BMI will be computed by dividing body mass (kg) by stature (m2).
Dietary intake | Baseline to 24 weeks
  To help interpret whether changes in body composition can be solely attributed to the PA intervention, dietary intake will also be assessed at the same time points as the other variables of interest. The participating parent or legal guardian will maintain a food record of the child's diet during two days of the week and one day on the weekend. In this record the parent will include quantity of food and fluids consumed, the preparation method, and the brand of the product. Before the baseline measurement, parents will attend a training session with a registered dietitian to learn how to estimate portion sizes and keep a food record. The information collected through the food records will be entered into The Food Processor, ESHA Research, Salem, OR, USA program and analyzed for macronutrient percent intake and total calories.
Parent confidence | Baseline to 24 weeks
  Parent's Confidence: will be measured by the Proxy Self-efficacy questionnaire (Shields CA, & Brawley LR. (2006) Preferring proxy-agency: Impact on self-efficacy for exercise. Journal of Health Psychology,11, 904-914) to assess parents' confidence and self-efficacy in scheduling and managing their child's physical activity behaviors and adherence to the physical activity program.
Parent influence | Baseline to 24 weeks
  Parent Influence: will be measured by the Parental Influence Question is Parental Social Control (Wilson, K.S., Spink, K.S., & Priebe, C.S. (2010). Parental social control in reaction to a hypothetical lapse in their child's activity: The role of parental activity and importance. Psychology of Sport and Exercise, 11, 231-237) to assess how the specific tactics parents choose to motivate their child influences the child's physical activity levels.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela A Rubin, Ph.D., Principal Investigator — California State University Fullerton, Department of Kinesiology
Locations (2):
- United States (2):
  - California State University Fullerton, Fullerton, California
  - University of Florida Gainesville, Gainesville, Florida

REFERENCES:
- [Derived] Rubin DA, Wilson KS, Castner DM, Dumont-Driscoll MC. Changes in Health-Related Outcomes in Youth With Obesity in Response to a Home-Based Parent-Led Physical Activity Program. J Adolesc Health. 2019 Sep;65(3):323-330. doi: 10.1016/j.jadohealth.2018.11.014. Epub 2019 Mar 2. PMID 30833118
- [Derived] Rubin DA, Wilson KS, Dumont-Driscoll M, Rose DJ. Effectiveness of a Parent-led Physical Activity Intervention in Youth with Obesity. Med Sci Sports Exerc. 2019 Apr;51(4):805-813. doi: 10.1249/MSS.0000000000001835. PMID 30407275
- [Derived] Rubin DA, Wilson KS, Honea KE, Castner DM, McGarrah JG, Rose DJ, Dumont-Driscoll M. An evaluation of the implementation of a parent-led, games-based physical activity intervention: the Active Play at Home quasi-randomized trial. Health Educ Res. 2019 Feb 1;34(1):98-112. doi: 10.1093/her/cyy035. PMID 30346530
- [Derived] Rubin DA, Wilson KS, Wiersma LD, Weiss JW, Rose DJ. Rationale and design of active play @ home: a parent-led physical activity program for children with and without disability. BMC Pediatr. 2014 Feb 14;14:41. doi: 10.1186/1471-2431-14-41. PMID 24529259